CLINICAL TRIAL: NCT06559111
Title: Postoperative Care After Operatively Treated Ankle Fractures With Cast or Functional Ankle Orthosis. A 2-year, Prospective, Randomized Clinical Trial
Brief Title: Cast or Functional Ankle Orthosis After Ankle Fracture Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Töölö Hospital (Other)
Collaborators: Tampere University Hospital (Other)
Responsible Party: Principal Investigator, Lasse Rämö, Orthopaedic Surgeon, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 06121917
Record Dates: First submitted 2024-08-14; First posted 2024-08-19 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Ankle Fracture; Postoperative Treatment
MeSH Terms: conditions — Ankle Fractures | interventions — Braces

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bracing group (Experimental): Participants in the bracing group had a cast for 2 weeks after the surgery followed by ankle brace for 4 weeks.
  Interventions: Device: 2-week casting followed by 4-week bracing
- Casting group (Active Comparator): Participants in the casting group had a cast for 6 weeks after the surgery.
  Interventions: Device: 6-week casting

INTERVENTIONS:
Device: 2-week casting followed by 4-week bracing — Participants in the bracing group had a cast for 2 weeks after the surgery followed by ankle brace for 4 weeks.
  Arms: Bracing group
Device: 6-week casting — Participants in the casting group had a cast for 6 weeks after the surgery.
  Arms: Casting group

SUMMARY:
The goal of this randomized clinical trial was to compare the effect of 6-week casting versus 2-week casting followed by 4-week ankle bracing in adult patients with surgically treated ankle fractures.

The primary outcome measures used were the functional results 3 months after surgery evaluated using two functional outcome measures (Olerud and Molander score and Kaikkonen score) and the patient return to work.

In the casting group, the traditional plaster was changed to a fiberglass one at 2 weeks and the cast treatment continued until 6 weeks. In the functional treatment group, the traditional plaster cast was changed to an reusable semi-rigid plastic orthosis (Aircast) at 2 weeks after surgery and its use was continued as an ankle support for up to 6 weeks. Follow-ups including subjective and objective evaluations were at 2, 6, 12 and 52 weeks and at 2 years postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Weber A or B type ankle fracture
* uni-, bi- or trimalleolar injury and/or fibular displacement of >2 mm in any plane on the radiographs

Exclusion Criteria:

* Weber C injury necessitating syndesmotic fixation
* Pilon injury
* Inadequate co-operation
* Other severe concomitant injuries

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 134 (Actual)
Dates: Start 2005-12-01 (Actual); Primary Completion 2010-06-16 (Actual); Study Completion 2012-03-16 (Actual)

PRIMARY OUTCOMES:
Olerud-Molander score | 3 months and 24 months
  Patient-reported outcome measure, 0-100 points, higher points indicating better result.

SECONDARY OUTCOMES:
Olerud-Molander score | 6 weeks and 12 months
  Patient-reported outcome measure, 0-100 points, higher points indicating better result.
Kaikkonen score | 6 weeks, 3, 12, and 24 months
  Patient-reported outcome measure, 0-100 points, higher points indicating better result.
Visual Analog Scale for Pain | 6 weeks, 3, 12, and 24 months
  0-10, higher score indicating more pain.
Swelling of the ankle | 6 weeks, 3, 12, and 24 months
  Circumference in millimetres compared to unaffected side
Atrophy of the calf muscles | 6 weeks, 3, 12, and 24 months
  Circumference in millimetres compared to unaffected side
Ankle active dorsiflexion | 6 weeks, 3, 12, and 24 months
  Degrees compared to unaffected side
Ankle active plantarflexion | 6 weeks, 3, 12, and 24 months
  Degrees compared to unaffected side
Return-to-work | Within 24 months
  Days after the injury
Subjective symptoms and return to activities | 2 and 6 weeks; 3, 12, and 24 months
  The patients were questioned about the subjective symptoms (pain, swelling, stiffness and giving way) and about the compliance of using the cast or brace. In addition the patients were asked about the length of their inability to work and participate in the daily activities and/or sports at the preinjury level.

OTHER OUTCOMES:
Complications | 2 and 6 weeks; 3, 12, and 24 months
  Infection, loss of reduction, implant loosening, deep vein thrombosis

CONTACTS AND LOCATIONS:
Overall Officials: Teppo Järvinen, Prof, Study Chair — Helsinki University Central Hospital

IPD SHARING:
Plan to Share IPD: No